CLINICAL TRIAL: NCT02587039
Title: An Intervention to Reduce Delirium After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Charles Brown, MD, Assistant Professor of Anesthesiology and Critical Care, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00030360
Record Dates: First submitted 2014-07-09; First posted 2015-10-27 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Delirium; Congenital Heart Disease; Coronary Artery Disease; Heart Valve Disease
Keywords: delirium; heart; valve; graft; surgery; coronary
MeSH Terms: conditions — Delirium; Heart Defects, Congenital; Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control: Usual care (Placebo Comparator): This group will receive usual care and delirium assessments.
  Interventions: Behavioral: Delirium Assessment
- Treatment: Ischemic Pre-conditioning (Experimental): Remote Ischemic pre-conditioning before cardiac surgery and delirium assessments.
  Interventions: Procedure: Remote ischemic pre-conditioning; Behavioral: Delirium Assessment

INTERVENTIONS:
Procedure: Remote ischemic pre-conditioning — Remote ischemic preconditioning is exposure to a brief period ischemia to an area or limb that is not involved in surgery. This intervention is believed to reduce the incidence of cerebral (brain) ischemia during cardiac surgery.
  Arms: Treatment: Ischemic Pre-conditioning
Behavioral: Delirium Assessment — The Delirium assessment consist of a validated psychiatric screening tool called the Confusion Assessment Method. We will use this tool to determine if patients have any confusion after surgery.

SUMMARY:
Patients that have cardiac surgery may suffer from unrecognized cerebral ischemia or loss of blood flow to the brain temporarily during surgery. This temporary loss of blood flow to the brain may result in a condition called delirium. Delirium is a type temporary confusion. There are some strategies that can help reduce cerebral ischemia during cardiac surgery which can help lead to a reduction in the incidence of delirium. The investigator believes that a strategy called remote ischemic preconditioning will help to reduce the incidence of delirium incidence after cardiac surgery.

Remote ischemic preconditioning is a brief exposure to ischemia. This brief exposure to ischemia occurs in an area of the body that is not undergoing a procedure. This brief exposure to ischemia is not long enough to cause any damage to the body and it has been demonstrated to help protect against more severe ischemic injury that may occur later during surgery. In this study the investigator will use remote ischemic preconditioning to see if it can reduce the incidence delirium after cardiac surgery.

DETAILED DESCRIPTION:
Delirium is common after cardiac surgery, occurring in 45-55% of patients, and is independently associated with increased postoperative complications, reduced functional capacity, cognitive decline, and increased mortality. Although the pathophysiology of delirium is unclear, a leading hypothesis is that delirium results from unrecognized cerebral ischemia during surgery. In preliminary data from the investigators group, delirium was reduced in patients randomized to optimal blood pressure control during cardiopulmonary bypass, using novel technology that determines an individual patient's lower limit of cerebral autoregulation. Thus, patients undergoing cardiac surgery may suffer from unrecognized cerebral ischemia that contributes to delirium, and strategies to attenuate the effects of cerebral ischemia may reduce the incidence of delirium.

Ischemic preconditioning represents a novel strategy to attenuate the effects of cerebral ischemia during cardiac surgery. Exposure to a brief period of ischemia, below the threshold for tissue injury, has been demonstrated to protect against the harmful effects of a subsequent more severe ischemic insult, in both animal and human studies. The protection provided by ischemic preconditioning may also be effective when the preconditioning is applied to a location remote from the organ of interest (i.e. a limb). Recently, a large randomized trial in patients undergoing cardiac surgery demonstrated a survival benefit among patients randomized to remote ischemic preconditioning vs. placebo. Remote ischemic preconditioning was achieved by simple inflation of a blood pressure cuff to supra-systolic pressures for 5 minutes, repeated for 3 cycles. However, neurological outcomes were not assessed in this trial, although animal models support potential neurological protection following remote ischemic preconditioning.

In this study the investigator will examine whether remote ischemic preconditioning can reduce delirium, functional decline, and biomarkers of cerebral injury after cardiac surgery. The investigator will explore the mechanism of preconditioning by examining proteomic analyses in a subset of patients. These results will provide data to support an NIH trial to examine the protective effects of remote ischemic preconditioning in cardiac surgery, identify potential mechanisms of action and potential targets for therapeutic pharmacologic interventions.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years old
* Undergoing coronary artery bypass and/or valve surgery

Exclusion Criteria:

* Mini mental state exam < 23
* Delirium at baseline
* Inability to speak and understand English
* Severe hearing impairment, resulting in inability to converse
* Planned use of intraoperative ketamine
* Inability to place or tolerate upper extremity tourniquet
* Hemoglobinopathy (e.g. sickle cell disease)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incident Delirium | First four postoperative days
  Delirium will be assessed using the Confusion Assessment Method (CAM) on three of the first four postoperative days. The primary outcome will be positive if delirium occurs by CAM criteria at any of these assessments

SECONDARY OUTCOMES:
Levels of novel cerebral injury biomarkers | Within 1 hour before the surgical incision, immediately after cardiopulmonary bypass, 2 hours after cardiopulmonary bypass, and 20 hours after skin closure
  Biomarkers include inflammatory proteins, and markers of neuronal damage or change in homeostasis, including glial fibrillary acidic protein and neurotrophic factors

OTHER OUTCOMES:
Instrumental Activities of Daily Living | 1 month and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Charles Brown, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Nakano M, Nomura Y, Suffredini G, Bush B, Tian J, Yamaguchi A, Walston J, Hasan R, Mandal K, Schena S, Hogue CW, Brown CH 4th. Functional Outcomes of Frail Patients After Cardiac Surgery: An Observational Study. Anesth Analg. 2020 Jun;130(6):1534-1544. doi: 10.1213/ANE.0000000000004786. PMID 32384343
- [Derived] Nomura Y, Nakano M, Bush B, Tian J, Yamaguchi A, Walston J, Hasan R, Zehr K, Mandal K, LaFlam A, Neufeld KJ, Kamath V, Hogue CW, Brown CH 4th. Observational Study Examining the Association of Baseline Frailty and Postcardiac Surgery Delirium and Cognitive Change. Anesth Analg. 2019 Aug;129(2):507-514. doi: 10.1213/ANE.0000000000003967. PMID 30540612